CLINICAL TRIAL: NCT01863667
Title: A Phase III, Multicenter, Double-Blind, Randomized Trial to Evaluate the Safety and Efficacy of MK-3102 Compared With Glimepiride in Subjects With Type 2 Diabetes Mellitus For Whom Metformin is Inappropriate Due to Intolerance or Contraindication
Brief Title: A Study to Evaluate the Safety and Efficacy of Omarigliptin (MK-3102) Compared With Glimepiride in Participants With Type 2 Diabetes Mellitus for Whom Metformin is Inappropriate (MK-3102-027)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3102-027; 2013-000301-23 (EudraCT Number)
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omarigliptin (Experimental): Participants receive an omarigliptin (MK-3102) 25 mg capsule once weekly and glimepiride placebo tablet(s) once daily, for 54 weeks.
  Interventions: Drug: Omarigliptin; Drug: Glimepiride Placebo
- Glimepiride (Active Comparator): Participants receive glimepiride 1 mg and/or 2 mg tablet(s) (maximum dose 6 mg/day) once daily and an omarigliptin placebo capsule once weekly, for 54 weeks.
  Interventions: Drug: Glimepiride; Drug: Omarigliptin Placebo

INTERVENTIONS:
Drug: Omarigliptin — Omarigliptin (MK-3102) 25 mg capsule administered orally once weekly
  Arms: Omarigliptin
Drug: Glimepiride — Glimepiride tablet 1 mg and/or 2 mg (uptitrated to a maximum dose 6 mg/day) administered orally once daily with breakfast or the first main meal
  Other Names: AMARYL®; GLIMY
  Arms: Glimepiride
Drug: Omarigliptin Placebo — Matching placebo to omarigliptin capsule administered orally once weekly
  Arms: Glimepiride
Drug: Glimepiride Placebo — Matching placebo to glimepiride tablet administered orally once daily with breakfast or the first main meal
  Arms: Omarigliptin

SUMMARY:
This trial will assess the safety and efficacy of omarigliptin (MK-3102) compared with the sulfonylurea, glimepiride, in type 2 diabetes mellitus participants who are metformin intolerant or who have a contraindication to the use of metformin. The primary hypothesis is that after 54 weeks, the mean change from baseline in hemoglobin A1c (A1C) in participants treated with omarigliptin is non-inferior compared with that in participants treated with glimepiride.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus
* Have intolerability to metformin ≥1000 mg/day or have a contraindication to the use of metformin
* Females of reproductive potential agree to remain abstinent or use or have their partner use 2 acceptable methods of birth control

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis or assessed by the investigator as possibly having type 1 diabetes
* Has been treated with:

  1. A thiazolidinedione (TZD) within 4 months of study participation, or
  2. A glucagon-like peptide-1 (GLP-1) receptor mimetic or agonist (such as exenatide or liraglutide) within 6 months of study participation, or
  3. Insulin within 12 weeks prior to study participation, or
  4. Dual antihyperglycemic agent (AHA) therapy within 12 weeks of study participation (4 months if a component of the dual AHA therapy was a TZD)
  5. Omarigliptin (MK-3102) at any time prior to study participation
* On a weight loss program and is not in the maintenance phase; has started a weight loss medication in the past 6 months; or has undergone bariatric surgery within 12 months prior to study participation
* Medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Human immunodeficiency virus (HIV)
* New or worsening coronary heart disease, congestive heart failure, myocardial infarction, unstable angina, coronary artery intervention, stroke or transient ischemic neurological disorder within the past 3 months
* History of malignancy ≤5 years prior to study participation except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* Clinically important hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* Pregnant or breast-feeding, or is expecting to conceive or donate eggs during the trial, including 21 days following the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-07-08 (Actual); Primary Completion 2014-04-03 (Actual); Study Completion 2014-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis Link — http://www.merck.com/clinical-trials/study.html?id=3102-027&kw=3102-027&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had a 1-week Screening Period; an oral antihyperglycemic agent (AHA) "wash-off" period of 8 weeks for participants on oral AHAs; a 2-week single-blind placebo run-in period; and a 54-week double-blind treatment period.
Groups:
- Omarigliptin: Participants received an omarigliptin (MK-3102) 25 mg capsule once weekly and glimepiride placebo tablet(s) once daily, for 54 weeks.
- Glimepiride: Participants received glimepiride 1 mg and/or 2 mg tablet(s) (maximum dose 6 mg/day) once daily and an omarigliptin placebo capsule once weekly, for 54 weeks.
Period: Overall Study
Arm/Group | Omarigliptin | Glimepiride
Started | 33 | 32
Completed | 0 | 0
Not Completed | 33 | 32
Not completed — Adverse Event | 1 | 0
Not completed — Study terminated by Sponsor | 30 | 30
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omarigliptin | Glimepiride | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (14.1) | 56.8 (9.9) | 57.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 54
Description: A1C is measured as a percent. Thus, this change from baseline reflects the Week 54 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 54
Population: Full Analysis Set defined as all participants who received at least one dose of study drug and had a baseline measurement or a post-randomization measurement. Due to the early termination of the study, no participants completed Week 54.
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is any untoward medical occurrence in a participant administered study drug which does not necessarily have a causal relationship with the treatment. Adverse events may include the onset of new illness and the exacerbation of pre-existing conditions.
Time Frame: Up to 57 weeks (including 3 weeks following the last dose of study drug)
Population: All participants as treated defined as all randomized participants who received at least one dose of study drug and were included in the treatment group corresponding to the study drug they actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 33 | 32
Percentage of participants | 9.1 | 15.6

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: as for outcome 2
Time Frame: Up to 54 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 33 | 32
Percentage of participants | 3 | 0

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 54
Description: This change from baseline reflects the FPG level at Week 54 minus the FPG level at Week 0.
Time Frame: Baseline and Week 54
Population: as for outcome 1
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants Achieving an A1C Goal <7.0% or <6.5% After 54 Weeks of Treatment
Description: Percentage of participants achieving glycemic goal (A1C <7% or <6.5%) after 54 weeks of treatment.
Time Frame: 54 weeks
Population: as for outcome 1
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants Meeting the Composite Endpoint of an A1C Decrease >0.5%, No Symptomatic Hypoglycemia, and No Body Weight Gain After 54 Weeks of Treatment
Description: Percentage of Participants who had an A1C decrease >0.5%, no symptomatic hypoglycemia, and no body weight gain after 54 weeks of treatment
Time Frame: 54 weeks
Population: as for outcome 1
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants With an Adverse Event of Symptomatic Hypoglycemia
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered study drug which does not necessarily have a causal relationship with the treatment. AEs may include the onset of new illness and the exacerbation of pre-existing conditions. Per protocol, an adverse event was defined as symptomatic hypoglycemia if hypoglycemia was an adverse event collected on the AE form AND the symptoms associated with it were collected on the hypoglycemia assessment (HA) form. Due to the early termination of the study, the HA form information was not assessed; therefore, this endpoint cannot be reported.
Time Frame: Up to 54 weeks
Population: as for outcome 2
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Body Weight at Week 54
Description: Body weight was to be measured (in duplicate) using a calibrated digital scale.
Time Frame: Baseline and Week 54
Population: All participants as treated defined as all randomized participants who received at least one dose of study drug and were included in the treatment group corresponding to the study drug they actually received. Due to the early termination of the study, no participants completed Week 54.
Arm/Group | Omarigliptin | Glimepiride
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 57 weeks (including 3 weeks following last dose of study drug)
Description: All participants as treated defined as all randomized participants who received at least one dose of study drug and were included in the treatment group corresponding to the study drug they actually received.
Arm/Group | Omarigliptin | Glimepiride
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (N=33) | Glimepiride (N=32)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated based on business decisions only, and not due to any unexpected safety or efficacy concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.